CLINICAL TRIAL: NCT05298046
Title: A Phase 1, Randomized, Placebo-Controlled, Double-Blind, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of TAVO101 in Adult Healthy Subjects
Brief Title: Study of TAVO101 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tavotek Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 59870001
Record Dates: First submitted 2021-12-29; First posted 2022-03-28 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- TAVO101: Low dose (Experimental): TAVO101: TAVO101 single ascending dose IV infusion.
  Interventions: Drug: Experimental: TAVO101
- TAVO101: Medium dose (Experimental): TAVO101: TAVO101 single ascending dose IV infusion.
  Interventions: Drug: Experimental: TAVO101
- TAVO101: High dose (Experimental): TAVO101: TAVO101 single ascending dose IV infusion.
  Interventions: Drug: Experimental: TAVO101
- Placebo (Placebo Comparator): Placebo single ascending dose IV infusion.
  Interventions: Other: Other: Placebo

INTERVENTIONS:
Drug: Experimental: TAVO101 — TAVO101 single ascending dose IV infusion.
  Other Names: TAVO101
  Arms: TAVO101: High dose; TAVO101: Low dose; TAVO101: Medium dose
Other: Other: Placebo — Placebo single ascending dose IV infusion.
  Arms: Placebo

SUMMARY:
This is a Phase 1, single ascending dose study designed to investigate TAVO101, administered as an IV infusion in healthy subjects. This study is designed to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of TAVO101.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, placebo-controlled, single ascending dose (SAD), single site study. Six subjects will be enrolled into each of the 7 dosing cohorts. Subjects will be randomized at a ratio of 2:1 to receive TAVO101 or placebo. Two sentinel subjects will be utilized (1 active:1 placebo) in each cohort in a manner designed to maintain the blind. Subjects will be evaluated for safety throughout the study up through day 196.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 and ≤ 65 years of age, inclusive.
* Subjects must have a body weight range of ≥50 kg and≤100 kg, inclusive, and BMI ≥ 18.0 and ≤ 30.0 kg/m2, inclusive at Screening and Day-1.
* Subjects must be healthy based on clinical laboratory tests performed at Screening and Day-1.
* Females of childbearing potential who are sexually active with a male partner must agree to use a highly effective method of contraception from Screening through 196 days after the final dose of study drug.
* Males who are sexually active and whose partners are females of childbearing potential must agree to use condoms from Screening through 196 days, after administration of the last dose of study drug and their partners must be willing to use a highly effective method of contraception from Screening through 196 days after the last dose of study drug.
* Males must agree to not donate sperm from Screening through 196 days, after the last dose of study drug administration.
* Subjects may be social smokers, defined as <5 cigarettes/month in last 6 months and must have negative cotinine test at Screening and check-in.
* Subjects will be considered eligible according to the following tuberculosis screening criteria's.
* Subjects must sign an Informed Consent Form.

Exclusion Criteria:

* Positive pregnancy test at Screening or baseline or is lactating.
* History or presence of conditions which, in the judgment of the investigator, are known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
* History or presence of conditions that may place the subject at increased risk as determined by the investigator.
* Subject has clinically significant laboratory abnormalities, or other clinically significant findings in the opinion of the investigator.
* Subject currently has or has had a history of any clinically significant medical illness or medical disorders the investigator considers should exclude the subject.
* Subject has a QT corrected according to Fridericia's formula (QTcF) interval >450 msec (for males) or >470 msec (for females), has a complete left or right bundle branch block, or has a history or current evidence of additional risk factors for Torsades de Pointes.
* History of surgery or major trauma within 16 weeks of Screening, or will not have fully recovered from surgery, or has surgery planned during the time the subject is expected to participate in the study, or within 17 weeks after the last dose of study drug administration.
* Subject plans to undergo non-major elective surgery within 5 weeks prior to study drug administration through EOS.
* Subject has a known or suspected intolerance or hypersensitivity to any components of the formulation of TAVO101 and its excipients used in this study.
* Subject has known hypersensitivity or severe allergies to food and or medication of clinical significance in the opinion of the investigator.
* History of alcohol abuse (i.e., more than 3 drinks per day), illicit drug use, physical dependence to any opioid, or any history of drug abuse or addiction within 12 months of Screening.
* Use of prescription medications (including hormone replacement therapy) within 14 days prior to administration of the study drug. By exception, prescription drugs, such as hormonal birth control, will be permitted.
* Use of over-the-counter drugs (including herbal preparations) within 7 days or 5 half-lives (if known), whichever is longer, prior to administration of the study drug.
* Has received a vaccination within 14 days prior to administration of the study drug.
* Has taken other investigational drugs or participated in any clinical study within 30 days or 5 half-lives (if known) of the investigational drug's PK, PD, or biological activity.
* Significant blood loss (>450mL) or has donated 1 or more units of blood or plasma within 6 weeks prior to study participation.
* Strenuous activity within 48 hours prior to CRU admission.
* Consumption of alcohol or caffeine-containing food or beverages within 48 hours prior to CRU admission.
* Positive urine drugs of abuse, alcohol, or cotinine screen.
* Positive test for HIV-1 or HIV-2 antibodies.
* Positive test for hepatitis B virus or hepatitis C virus consistent with current infection.
* Subject has liver function tests> 1.5x upper limit of normal (i.e., AST, ALT).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
The severity of adverse effects according to the National Cancer Institute's Common Terminology Criteria for AEs, Version 5.0 [Time Frame: Day 1 through Day 196] | 196 days
  To investigate the safety and tolerability of TAVO101 in healthy volunteers.
Changes in vital signs including oral temperature or tympanic temperature (C°) [Time Frame: Day 1 through Day 196] | 196 days
  To investigate the safety and tolerability of TAVO101 in healthy volunteers.
Changes in vital signs including respiratory rate (breaths per minute) [Time Frame: Day 1 through Day 196] | 196 days
  To investigate the safety and tolerability of TAVO101 in healthy volunteers.
Changes in vital signs including systolic and diastolic blood pressure (mmHg) [Time Frame: Day 1 through Day 196] | 196 days
  To investigate the safety and tolerability of TAVO101 in healthy volunteers.
Changes in vital signs including pulse rate (beats per minute) [Time Frame: Day 1 through Day 196] | 196 days
  To investigate the safety and tolerability of TAVO101 in healthy volunteers.

SECONDARY OUTCOMES:
Immunogenicity of TAVO101 [ Time Frame: Day 1 through Day 196 ] | 196 days
  Incidence of anti-drug antibodies (ADA) following dosing of TAVO101
Cmax (Maximum observed serum concentration ) [ Time Frame: Day 1 through Day 196 ] | 196 days
  To investigate the pharmacokinetics of TAVO101 in healthy volunteers.
tmax (time that Cmax was observed) [ Time Frame: Day 1 through Day 196 ] | 196 days
  To investigate the pharmacokinetics of TAVO101 in healthy volunteers.
AUC-last (Area under the serum concentration-time curve from time 0 to the time of the last quantifiable concentration; calculated using the linear/log trapezoid rule) [ Time Frame: Day 1 through Day 196 ] | 196 days
  To investigate the pharmacokinetics of TAVO101 in healthy volunteers.
AUC-inf (Area under the serum concentration-time curve from time 0 extrapolated to infinity) [ Time Frame: Day 1 through Day 196 ] | 196 days
  To investigate the pharmacokinetics of TAVO101 in healthy volunteers.
AUC0-t (Area under the serum concentration-time curve from time 0 to time t) [ Time Frame: Day 1 through Day 196 ] | 196 days
  To investigate the pharmacokinetics of TAVO101 in healthy volunteers.
t½ (Terminal elimination half-life) [ Time Frame: Day 1 through Day 196 ] | 196 days
  To investigate the pharmacokinetics of TAVO101 in healthy volunteers.
λz (Terminal elimination rate constant) [ Time Frame: Day 1 through Day 196 ] | 196 days
  To investigate the pharmacokinetics of TAVO101 in healthy volunteers.
CL (Systemic clearance) [ Time Frame: Day 1 through Day 196 ] | 196 days
  To investigate the pharmacokinetics of TAVO101 in healthy volunteers.
Vd (Volume of distribution) [ Time Frame: Day 1 through Day 196 ] | 196 days
  To investigate the pharmacokinetics of TAVO101 in healthy volunteers.

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No